CLINICAL TRIAL: NCT00004105
Title: A Phase I/II Study of Paclitaxel, Estramustine Phosphate, and Vinorelbine (PaclEVin)
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067324; P30CA016087 (NIH); NYU-9712; NCI-G99-1596
Record Dates: First submitted 1999-12-10; First posted 2004-05-25 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia; Lymphoma; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; unspecified adult solid tumor, protocol specific; childhood fibrosarcoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Sarcoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Fibrosarcoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Estramustine; Paclitaxel; Vinorelbine

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel
Drug: vinorelbine ditartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of vinorelbine, paclitaxel, and estramustine in treating patients who have advanced cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Establish the maximum tolerated doses (MTDs) and recommended Phase II doses (RPTDs) of vinorelbine and paclitaxel when combined with a fixed dose of estramustine in patients with advanced cancers or metastatic prostate cancer. II. Determine the toxicity pattern of this regimen at the MTDs and at the RPTDs in these patients. III. Make preliminary observations of antitumor activity in these patients treated with this regimen as leads for the Phase II portion of this study. IV. Establish the efficacy of the RPTDs of vinorelbine and paclitaxel when combined with estramustine in patients with prostate cancer who fulfill the criteria for the Phase II portion of this study.

OUTLINE: This is a dose escalation, multicenter study of vinorelbine and paclitaxel. Patients receive oral estramustine every 8 hours on days 0-2 and 7-9 and vinorelbine IV over 6-10 minutes immediately followed by paclitaxel IV over 1 hour on days 2 and 9. Courses repeat every 21 days. Patients with complete response, partial response, or stable disease continue treatment indefinitely in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of vinorelbine and paclitaxel until the maximum tolerated dose (MTD) of each drug is determined. The MTD is defined as the lowest dose at which 2 or more of 3-6 patients experience dose limiting toxicity. The recommended Phase II dose of vinorelbine or paclitaxel is defined as the dose immediately preceding the MTD.

PROJECTED ACCRUAL: A minimum of 12-16 patients will be accrued over 1 year for Phase I of the study and a total of 14-25 patients will be accrued for Phase II of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Phase I: Histologically proven advanced cancer that has failed or is not amenable to standard treatment Phase II: Histologically proven metastatic prostate cancer as documented by bone scan and rising PSA Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 0-2 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin greater than 9 g/dL (transfusion allowed) Hepatic: AST and ALT no greater than 4 times upper limit of normal Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No myocardial infarction within the past year No New York Heart Association class III or IV heart disease No uncontrolled cardiac dysrhythmia No angina pectoris No uncontrolled hypertension No cardiomyopathy Neurologic: No prior neuropathy No preexisting neurotoxicity Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Phase I: No prior vinorelbine (any schedule) or paclitaxel on a 24 hour or longer schedule At least 2 weeks since prior chemotherapy Phase II: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No radiotherapy to greater than 25% of bone marrow At least 3 weeks since prior radiotherapy No concurrent radiotherapy during courses 1 and 2. Surgery: No concurrent oncologic surgery during courses 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States